CLINICAL TRIAL: NCT05368610
Title: Effect of Very High Power-short Duration Ablation on Lesion Contiguity in Pulmonary Vein Isolation as Assessed by Late Gadolinium Enhancement Cardiovascular Magnetic Resonance
Brief Title: Lesion Contiguity in Very High Power-short Duration Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Till F. Althoff, Staff, Arrhythmia Section, Department of Cardiology, Hospital Clinic de Barcelona, University of Barcelona
Other Study IDs: QDOT-MRI
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Very high power-short duration ablation: PVI performed by point-by-point very high power-short duration radiofrequency ablation (QDOT-micro catheter, Biosense Webster; Qmode+; 90 W; 4 sec; target intertag distances: posterior wall 4 mm, proximity of the esophagus 5 mm, all other 3 mm)
- Matched control group conventional ablation: PVI performed by conventional point-by-point radiofrequency ablation (40 W; ablation index-guided: posterior wall 350, other 450; target intertag distance 3.0 - 5.0 mm)

SUMMARY:
This observational trial investigates the effect of very high power-short duration radiofrequency ablation on lesion contiguity as assessed by late gadolinium enhancement cardiovascular magnetic resonance (LGE-CMR). Patients with paroxysmal or early persistent atrial fibrillation (AF) scheduled for pulmonary vein isolation (PVI) undergo point-by-point ablation using the QDOT micro catheter applying Qmode+ (90W over 4 seconds). All patients receive an LGE-CMR 3 months after the procedure for ablation lesion assessment. Contiguity of LGE-CMR-detected ablation lesions will be compared with a matched control group of patients that have undergone PVI accomplished by ablation index-guided ablation with 40 W following the CLOSE protocol.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal or early persistent (max. 3 months) atrial fibrillation
* scheduled for PVI-only catheter ablation

Exclusion Criteria:

* long-standing persistent atrial fibrillation
* previous left atrial ablation
* claustrophobia preventing CMR
* sever renal insufficiency (GFR >30 ml/min)
* gadolinium contrast allergy
* presence of implantable devices not compatible with magnetic resonance
* pregnancy and lactation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for PVI-only catheter ablation at Hospital Clinic, University of Barcelona
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Ablation lesion contiguity as assessed by LGE-CMR | LGE-CMR at 3 months post-ablation
  Proportion of the circumferential ablation line covered by LGE (%)

CONTACTS AND LOCATIONS:
Overall Officials: Till F. Althoff, M.D., Principal Investigator — Hospital Clinic, University of Barcelona
Locations (1):
- Hospital Clinic, University of Barcelona, Barcelona, Catalonia, Spain